CLINICAL TRIAL: NCT01830790
Title: Effects of Sildenafil on Choroidal Thickness in Age-Related Macular Degeneration
Brief Title: Effects of Sildenafil on Choroidal Thickness in AMD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate support to complete recruitment/data analysis.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00042897
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Results first posted 2015-05-14 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-04

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Controls (Active Comparator): Healthy individuals >65 years old without ocular disease, who will be given a single dose of 100mg sildenafil citrate, then imaged with EDI-OCT to determine a change in choroidal thickness
  Interventions: Drug: Sildenafil citrate
- AMD patients (Experimental): Age-related macular degeneration (AMD) patients >65 years old without other ocular disease, who will be given a single dose of 100mg sildenafil citrate, then imaged with EDI-OCT to determine a change in choroidal thickness
  Interventions: Drug: Sildenafil citrate

INTERVENTIONS:
Drug: Sildenafil citrate — Single dose of 100mg Sildenafil citrate
  Other Names: Viagra; Revatio

SUMMARY:
Choroidal thinning has been hypothesized to partake in the pathogenesis of age-related macular degeneration (AMD), but it is not known if increasing choroidal thickness may potentially alter the disease course. Past studies have shown that a single dose of the phosphodiesterase type-5 inhibitor sildenafil citrate can increase choroidal thickness in young healthy patients. The investigators hypothesize that sildenafil may also increase choroidal thickness in eyes with AMD and perhaps potentially reduce AMD progression. Alternatively, if sildenafil has minimal effect on choroidal thickness in eyes in patients with AMD, such results may suggest that choroidal vascular compliance or stiffness is reduced in this condition. Patients seen at the Duke Eye Center with a diagnosis of AMD or age-matched control subjects with no macular pathology will be administered a single 100mg oral dose of sildenafil citrate (Viagra®; Pfizer), and undergo EDI-OCT imaging before and after treatment. Images obtained will be used to measure choroidal thickness, as well as central macular thickness (CMT) and macular volume (MV). Choroidal thickness changes after a single-dose sildenafil treatment in AMD patients will be compared with age-matched control subjects using standard statistical methods. By also correlating choroidal thickness changes with functional (visual acuity) and anatomical (CMT & MV) changes, the investigators hope to further their understanding of the choroid's role in aging and AMD pathogenesis. The safety of a single dose of sildenafil citrate will be addressed by excluding any patients with risk factors or using medications that are contraindicated for sildenafil as determined by careful informed consent and a study questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* has been diagnosed with AMD (362.50-52) or healthy controls as detailed above
* at least 65 years of age
* capable and willing to provide consent

Exclusion Criteria:

* History of previous photodynamic therapy (PDT), intravitreal corticosteroid injection, macular focal laser photocoagulation, panretinal photocoagulation, ocular ionizing irradiation, transpupillary thermotherapy, or any vitreoretinal surgeries
* History of central serous chorioretinopathy, polypoidal choroidal vasculopathy, uveitis, or diabetic retinopathy
* History of amblyopia, glaucoma, retinal detachment, retinal dystrophy, ocular trauma, ocular tumor, proliferative retinopathy, or epiretinal membrane with distortion of central macula
* History of myopia of more than 6 diopters (D) spherical equivalent
* History of uncontrolled diabetes or hypertension
* Current use of oral phosphodiesterase type 5 inhibitors (including sildenafil, avanafil, lodenafil, mirodenafil, tadalafil, vardenafil, udenafil, zaprinast)
* Current use of systemic corticosteroids
* Any contraindication to sildenafil use, including history of cardiovascular disease or stroke, hepatic cirrhosis (Child-Pugh A and B), severe renal impairment (creatinine clearance <30mL/min), anatomical deformation of the penis (such as angulation, cavernosal fibrosis, or Peyronie's disease), disorders predisposing to priapism (e.g. sickle cell anemia, multiple myeloma, or leukemia), or current use of organic nitrates, alpha-blockers, or potent cytochrome P450 3A4 inhibitors

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Fekrat, MD, Principal Investigator — Duke University Eye Center
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Controls | AMD Patients
Started | 0 | 10
Completed | 0 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | AMD Patients | Total
Number analyzed (Participants) | 0 | 10 | 10
Age, Categorical [Number; unit: participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 2 | 2
  >=65 years |  | 8 | 8
Gender [Number; unit: participants]
  Female |  | 4 | 4
  Male |  | 6 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Choroidal Thickness as Assessed on Enhanced-Depth Imaging Optical Coherence Tomography (EDI-OCT)
Time Frame: Baseline, 1 hour, and 3 hours post-treatment
Population: Study was terminated early due to inadequate support to complete recruitment/data analysis. No outcome measure data was collected.
Arm/Group | Healthy Controls | AMD Patients
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Central Foveal Thickness as Assessed by Optical Coherence Tomography (OCT)
Time Frame: Baseline, 1hour, and 3 hours post-treatment
Population: as for outcome 1
Arm/Group | Healthy Controls | AMD Patients
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Healthy Controls | AMD Patients
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/10
Other Adverse Events (participants affected / at risk) | 0/0 | 0/10

LIMITATIONS AND CAVEATS:
Study was terminated early due to inadequate support to complete recruitment/data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes